CLINICAL TRIAL: NCT05043233
Title: The Observation Study of Graves' Disease Cohort
Brief Title: Observation in the Treatment of Graves' Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Clinical Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 132563
Record Dates: First submitted 2021-08-30; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Patient Acceptance of Health Care
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — In the study, peripheral venous blood samples form paitents at 3 time points during follow-up(untreated, euthyorid status, and TRAb-neative status). Collection requirements: about 10ml venous blood should be collected by anticoagulant vacuum negative pressure blood collection vessel while the patient does not need to be fasting. Then their clinical parameters, including thyrotropin (TSH), free T3 (FT3), free T4 (FT4), thyroperoxidase antibody (TPOAb), thyroglobulin antibody (TgAb) and thyrotropin receptor antibody (TRAb) levels, thyroid-stimulating immunoglobulin (TSI) were measured by routine clinical laboratory methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Graves' disease: Graves' disease was diagnosed based on clinical symptoms and laboratory findings. The clinical symptoms included heat intolerance, fatigue, increased appetite, increased sweating, weight loss, muscle weakness, tremors, and diffusely enlarged thyroid glands. The laboratory results included increased serum concentrations of free thyroxine (FT4) and/ or free triiodothyronine (FT3), decreased basal thyroid-stimulating hormone (TSH) level, and TRAb positivity. All participants in this study would be treated with anti-thyroid drugs(MMI: methimazole) according to the 2016 ATA guildline.
  Interventions: Drug: Methimazole(MMI)

INTERVENTIONS:
Drug: Methimazole(MMI) — Methimazole is a widely used antithyroid drug and is often used in the treatment of Graves' disease hyperthyroidism

SUMMARY:
At present, there are still few observational studies on Graves' disease in China, and there are few research reports in this regard. In order to further carry out high-quality observational follow-up research on Graves' disease hyperthyroidism, including establishing standard diagnosis and treatment procedures, providing data support for the establishment of research protocols such as sample size and follow-up time estimation, this study was conducted at Ruijin Hospital, Shanghai Jiaotong University School of Medicine. The endocrinology clinic carried out the registration follow-up study of Graves' disease.

DETAILED DESCRIPTION:
Graves' disease is the main cause of clinically hyperthyroidism, accounting for about 75% to 80%, and it occurs in women of childbearing age. Clinical manifestations include: high eating, weight loss, sweating, palpitations, emotional excitement and other high metabolism Syndrome. Some patients may have manifestations such as infiltrating exophthalmos and pretibial mucinous edema.

Graves' disease is an organ-specific autoimmune disease characterized by the production of a specific antibody TRAb against thyroid stimulating hormone receptor (TSHR). TRAb can mimic the role of thyroid stimulating hormone, combined with TSHR, stimulating TRAb can cause continuous activation of cAMP, resulting in increased production and release of thyroid hormone. Excessive thyroid hormones in the circulation act on body tissues to cause hypermetabolism and goiter. The pathogenesis of Graves' disease is currently unclear. The three major factors of genetics, environment and immunity are involved in the onset of Graves' disease. There is no doubt that the immune factor is an important factor in the pathogenesis of Graves' disease hyperthyroidism. Studies have shown that CD4+ T cells play an important role in Graves disease. CD4+ T lymphocytes can accept antigens presented by antigen presenting cells, secrete cytokines and assist B lymphocytes to differentiate into plasma cells and produce antibodies. CD4+T accounts for about 40% to 60% of peripheral T cells and can be differentiated into various T cell subsets such as Th1, Th2, Th17, Th22, Th9 and Treg cells. Treg cells are regulatory T cells, mainly involved in the negative regulation of inflammation. Recent researches suggest that the decrease in Treg cell number or loss of function is related to the pathogenesis of various autoimmune diseases. The investigators' previous study showed that the proportion of Treg cells in peripheral blood mononuclear cell of patients with initial Graves' disease was significantly lower than that of healthy controls, and it was negatively correlated with TRAb levels. At the same time, studies have shown that in the early stage of Graves' disease, the number of pDC cells as the main antigen presenting cells has increased. In vitro studies have confirmed that pDC secretes IFN-α to induce differentiation of naive T cells and interferes with the normal immunosuppression of Treg cells. Function, induce apoptosis of Treg cells. Therefore, the weakened immunosuppressive effect of Treg cells also plays a role in the pathogenesis of Graves' disease.

Graves' disease is an autoimmune disease, but the current treatments for Graves' disease: antithyroid drugs, radioactive 131I, surgery, but there is no treatment method through direct immune modulation. Surgery and radioactive 131I treatment achieve rapid cure by removing or damaging the thyroid gland. Surgery is invasive treatment. There are neurovascular injury and anesthesia complications. Most patients with secondary thyroid dysfunction after radioactive 131I treatment require oral L-T4 for life.Compared with the other two methods, antithyroid drug treatment has the advantages of non-invasiveness, convenience, and ease of acceptance by patients, but it has the problems of long treatment duration, low remission rate, and easy recurrence. It also has the induction of agranulocytosis, liver function damage, and rash.

However, there are still few observational follow-up studies on Graves' disease in China, and there are few research reports in this regard.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-70 years old with normal BMI (18-25), who are diagnosed with Graves' disease hyperthyroidism in accordance with the 2016 American Thyroid Association's guidance at the first diagnosis, or patients who relapse after more than one year of medication withdrawal.

1. High metabolic symptoms such as fear of heat, sweating, and palpitations;
2. Diffuse enlargement of thyroid gland, B-ultrasound of thyroid gland indicates diffuse thyroid disease and increased blood flow of thyroid;
3. Serological detection of TSH levels decreased and FT3 and/or FT4 increased; meanwhile, TRAb was positive (TRAb>1.75 IU/L);
4. Accompanied by thyroid infiltrating ocular signs or pretibial mucous edema.

Exclusion Criteria:

1. Patients with Graves' disease who have previously undergone radioactive iodine 131 or surgery;
2. Blood routine WBC<3×109/L, neutrophils<1.5×109/L, or accompanied by other malignant blood diseases;
3. Patients with other serious heart, liver, lung, kidney disease or malignant tumors;
4. In the past six months, there is a history of using immunosuppressants or other autoimmune diseases such as systemic lupus erythematosus, Sjogren's syndrome, etc.;
5. Pregnant and lactating women; Allergies to the drugs used in the treatment plan; and any situation (medical, psychological, social, or geographical factors) that may endanger the safety of the patient or prevent the patient from successfully participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research object comes from the outpatients of Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine. The recruitment site is the Department of Endocrinology of Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
change in TRAb level (IU/L) | 12 weeks
Predict the risk of recurrence before the start of antithyroid drug therapy | through study completion, an average of 1 year

SECONDARY OUTCOMES:
change in FT3 level (pmol/L) | 12 weeks
change in FT4 level (pmol/L) | 12 weeks
change in TSH level (uIUm/L) | 12 weeks
change in TSI level (IU/L) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, MD,PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No